CLINICAL TRIAL: NCT02439606
Title: GlideRite® Rigid Stylet Versus Parker Flex-It Stylet for Orotracheal Intubation by GlideScope
Brief Title: GlideRite® Rigid Stylet Versus Parker Flex-It Stylet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Ashraf Arafat Abdelhalim, Assistant professor, Department of Anesthesia, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E-14-1074
Record Dates: First submitted 2015-04-01; First posted 2015-05-12 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Anesthesia
Keywords: GlideRite; Stylet; Parker; orotracheal; intubation; GlideScope

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glide Rite Rigid Stylet group (Active Comparator): Intubation with the GlideScope® video-laryngoscope and styletted the tracheal tube using manufacturer's GlideRite Rigid Stylet (GRS) (GVL - ST1; Verathon Medical Inc., Bothell, WA, USA). Time till successful intubation of the patient is calculated.
  Interventions: Device: Glide Rite Rigid Stylet group
- Parker-Flex-It Directional Stylet group (Experimental): Intubated with the GlideScope® video-laryngoscope and styletted the tracheal tube using Parker-Flex-It Directional Stylet (Parker Medical, Colorado, USA) (Flexi-Stylet). Time till successful intubation of the patient is calculated.
  Interventions: Device: Parker Flex-It directional stylet group

INTERVENTIONS:
Device: Glide Rite Rigid Stylet group — Intubation with the GlideScope® video-laryngoscope and styletted the tracheal tube using manufacturer's GlideRite Rigid Stylet (GRS) (GVL - ST1; Verathon Medical Inc., Bothell, WA, USA). Time till successful intubation of the patient is calculated.
  Arms: Glide Rite Rigid Stylet group
Device: Parker Flex-It directional stylet group — Intubated with the GlideScope® video-laryngoscope and styletted the tracheal tube using Parker-Flex-It directional Stylet (Parker Medical, Colorado, USA) (Flexi-Stylet). Time till successful intubation of the patient is calculated.
  Arms: Parker-Flex-It Directional Stylet group

SUMMARY:
This prospective randomized trial evaluated Parker Flex-It stylet as an alternative to manufacturer, s GlideRite® Rigid Stylet to aid intubation with the GlideScope in patients undergoing elective non-cardiac surgery that required general anesthesia with orotracheal intubation.

DETAILED DESCRIPTION:
The GlideScope® Ranger (GVL; Verathon Medical Inc., Bothell, WA, USA) is a novel portable, reusable video laryngoscope that has provided superior laryngeal visualization to facilitate tracheal intubation especially in the management of difficult airways; it provides indirect visualization of the glottis with a pronounced angle of 60° in the blade. It has separate monitor connected to the handle via a cable. The tip of the blade is equipped with high-resolution digital video camera, an LED light and an antifogging system.

Unlike the Macintosh laryngoscope, an indirect laryngoscope such as the GlideScope device provides a view of the glottis without the need to align the oral pharyngeal and laryngeal axes facilitating an excellent glottic visualization. However, insertion and advancement of the endotracheal tube (ETT) may be more difficult to pass through the vocal cords than direct laryngoscopy, and trauma is possible.

The GlideScope have shown to function better when used in conjunction with use of a stylet to guide insertion of endotracheal tube. The GlideRite Rigid Stylet (GRS) is a reusable rigid steel stylet, specifically designed by the manufacturer to resemble the distal part of the GVL blade for clear view of the airway, enabling quick intubation , its curvature approaches 90° with a radius of curvature of approximately 6 cm.

Various investigators have recommended different curvatures of the ETT/stylet to optimally direct it into the trachea, including matching the blade's 60° angle, configuring the ETT with a 90° bend, or using a J-shaped ETT. Other potential strategies may include the use of a flexible stylet that allows active modification of the tip of the tracheal tube during use.

The Parker Flex-It Directional Stylet (FIS, Parker Medical, Highlands Ranch, CO) is a 2-piece plastic stylet, can be used for oral intubation, and allows continuous adjustment of the tube curvature during an intubation to enable the tube to follow the curvature of the airway. We hypothesized that the use of Parker Flex-It stylet to guide ETT might offer some benefit over the GRS.

Therefore, the purpose of this study was to determine the optimal stylet-tracheal tube strategy for use with the GlideScope® laryngoscope. We compared efficacy of the two intubating aids including GlideRite® Rigid Stylet versus Parker Flex-It stylet for orotracheal intubation in terms of the total intubation time (primary outcome), ease of intubation, the number of intubation attempts , the number of optimization man oeuvres and possible trauma (secondary outcomes) when used by experienced GlideScope operators.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I&II,
* body mass index (BMI) < 35
* elective non-cardiac surgery
* general anaesthesia with orotracheal intubation

Exclusion Criteria:

* Anticipated difficult airway,
* need for rapid sequence induction,
* ASA physical status III-V,
* increase risk of gastric aspiration such as gastro- oesophageal reflux,
* pregnancy,
* patients who had no teeth, loose teeth or oral trauma, known pathology or previous surgery to the mouth, pharynx, larynx or cervical spine and any reason why the GlideScope is not, or could not be used.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2014-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
total intubation time | measured during intubation ( up to 120 seconds)
  the time from insertion of the blade of the GlideScope into the oral airway to the appearance of end-tidal carbon dioxide (ETCO2) curve of at least 30 mmHg on the anesthesia monitor after insertion of the tracheal tube.

SECONDARY OUTCOMES:
number of intubation attempts before successful intubation | 5minutes

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf Abdelhalim, MD, Principal Investigator — King Saud University